CLINICAL TRIAL: NCT02093039
Title: Informed Decision Users of the Health System and Participation in Organized Screening for Breast Cancer : a Qualitative Analysis
Brief Title: Informed Decision Users of the Health System and Participation in Organized Screening for Breast Cancer
Acronym: DECIDEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-01
Record Dates: First submitted 2014-03-19; First posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-03

CONDITIONS: Healthy; Breast Cancer
Keywords: breast cancer screening; patient decision aids; informed decision; empowerment; randomized control trial; From 50 to 74 years old; invited to national breast cancer screening
MeSH Terms: conditions — Breast Neoplasms; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Decision aid group (Experimental): Women allocated to the decision aid group received an invitation to participate in the national breast cancer screening program and the specially-designed decision aid (a leaflet), by mail.
  Interventions: Device: decision aid group
- Control group (No Intervention): Women in the control group received an invitation and the usual standard information by mail.

INTERVENTIONS:
Device: decision aid group — The paper-based leaflet DECIDEO is a 12-page pocket leaflet providing scientific information about the advantages and disadvantages of participating in the national breast screening program, understandable by all, constructed to conform with the International Patient Decision Aid Standards
  Arms: Decision aid group

SUMMARY:
The aim of this study is to assess the impact of a decision aid leaflet on the participation of women invited to participate in the French national breast cancer screening program.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged between 50 and 74 years old living in 11 French departments

Exclusion Criteria:

-

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16000 (Actual)
Dates: Start 2009-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
women's attendance rate for the breast cancer screening program during the 12 months following the invitation | 12 months

SECONDARY OUTCOMES:
the delay between the invitation and the date of attendance for breast cancer screening | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Franck CHAUVIN, MDPhD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

REFERENCES:
- [Background] Bray F, Ren JS, Masuyer E, Ferlay J. Global estimates of cancer prevalence for 27 sites in the adult population in 2008. Int J Cancer. 2013 Mar 1;132(5):1133-45. doi: 10.1002/ijc.27711. Epub 2012 Jul 26. PMID 22752881
- [Background] Olsson S, Andersson I, Karlberg I, Bjurstam N, Frodis E, Hakansson S. Implementation of service screening with mammography in Sweden: from pilot study to nationwide programme. J Med Screen. 2000;7(1):14-8. doi: 10.1136/jms.7.1.14. PMID 10807141
- [Background] Walter LC, Lewis CL. Maximizing informed cancer screening decisions. Arch Intern Med. 2007 Oct 22;167(19):2027-8. doi: 10.1001/archinte.167.19.2027. No abstract available. PMID 17954794
- [Background] Raffle AE. Informed participation in screening is essential. BMJ. 1997 Jun 14;314(7096):1762-3. doi: 10.1136/bmj.314.7096.1762a. No abstract available. PMID 9202520
- [Background] Barratt A, Trevena L, Davey HM, McCaffery K. Use of decision aids to support informed choices about screening. BMJ. 2004 Aug 28;329(7464):507-10. doi: 10.1136/bmj.329.7464.507. PMID 15331483
- [Background] Elwyn G, O'Connor A, Stacey D, Volk R, Edwards A, Coulter A, Thomson R, Barratt A, Barry M, Bernstein S, Butow P, Clarke A, Entwistle V, Feldman-Stewart D, Holmes-Rovner M, Llewellyn-Thomas H, Moumjid N, Mulley A, Ruland C, Sepucha K, Sykes A, Whelan T; International Patient Decision Aids Standards (IPDAS) Collaboration. Developing a quality criteria framework for patient decision aids: online international Delphi consensus process. BMJ. 2006 Aug 26;333(7565):417. doi: 10.1136/bmj.38926.629329.AE. Epub 2006 Aug 14. PMID 16908462
- [Background] Mathieu E, Barratt A, Davey HM, McGeechan K, Howard K, Houssami N. Informed choice in mammography screening: a randomized trial of a decision aid for 70-year-old women. Arch Intern Med. 2007 Oct 22;167(19):2039-46. doi: 10.1001/archinte.167.19.2039. PMID 17954796
- [Background] Edwards A, Unigwe S, Elwyn G, Hood K. Effects of communicating individual risks in screening programmes: Cochrane systematic review. BMJ. 2003 Sep 27;327(7417):703-9. doi: 10.1136/bmj.327.7417.703. PMID 14512475